CLINICAL TRIAL: NCT02286843
Title: Can HER2 Targeted PET/CT Imaging Identify Unsuspected HER2 Positive Breast Cancer Metastases, Which Are Amenable to HER2 Targeted Therapy?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-156
Record Dates: First submitted 2014-11-06; First posted 2014-11-10 (Estimated); Results first posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2020-07

CONDITIONS: Breast Cancer Metastases; HER2 Positive Breast
Keywords: 89Zr-trastuzumab; PET/CT; 14-156; 89Zr-pertuzumab; HER2-targeted
MeSH Terms: interventions — zirconium-89-trastuzumab; Positron Emission Tomography Computed Tomography

ARMS (1):
- HER2-targeted PET/CT (Experimental): Pts with confirmed HER2- breast cancer will then undergo HER2-targeted PET/CT. 89Zr-trastuzumab is a novel radiotracer which allows excellent visualization of HER2+ lesions. 89Zr-pertuzumab is a novel radiotracer which may allow for specific visualization of HER2+ lesions. PET/CT imaging with these novel radiotracers will allow evaluation of all identifiable malignant lesions, rather than evaluation of only single lesions by biopsy. Avid lesions will be considered suspicious for HER2+ malignancy. Pts with at least one 89Zr-trastuzumab or 89Zr-pertuzumab avid lesion will be biopsied to confirm HER2+ pathology. From these 50 pts, we will determine the proportion of HER2- primary breast cancer pts that express HER2+ malignancy imagable by HER2-targeted PET/CT. Pts recruited to the protocol, but then drop out prior to HER2-targeted PET/CT due HER2+ disease being identified on retesting of the patient's archived tissue samples, will be replaced with newly recruited pts.
  Interventions: Radiation: 89Zr-trastuzumab; Device: PET/CT scan; Radiation: 89Zr-pertuzumab

INTERVENTIONS:
Radiation: 89Zr-trastuzumab
Device: PET/CT scan
Radiation: 89Zr-pertuzumab

SUMMARY:
Some breast cancer cells make a protein called Human Epidermal Growth factor receptor 2 (HER2). Patients with HER2 positive (HER2+) breast cancer receive medicine that attacks HER2, which helps these patients live longer. Some HER2 negative (HER2-) breast cancer patients also benefit from medicines that attack HER2, but we do not know why or which patients will benefit. This study uses a new imaging method, HER2-targeted PET/CT, to identify patients that may benefit from medicines that attack HER2. This is experimental.

ELIGIBILITY:
Inclusion Criteria:

* Women age > 18
* Biopsy proven HER2 negative primary breast cancer and biopsy proven metastatic disease.
* 5 or more foci of demonstrable metastases on recent imaging modalities (CT, MR, FDG PET/CT)
* ECOG performance score of 0-2

Exclusion Criteria:

* Life expectancy < 3months
* Pregnancy or lactation
* Patients who cannot undergo PET/CT scanning because of weight limits
* CNS only disease on recent imaging

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2014-11-06 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Ulaner, MD,PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Ulaner GA, Carrasquillo JA, Riedl CC, Yeh R, Hatzoglou V, Ross DS, Jhaveri K, Chandarlapaty S, Hyman DM, Zeglis BM, Lyashchenko SK, Lewis JS. Identification of HER2-Positive Metastases in Patients with HER2-Negative Primary Breast Cancer by Using HER2-targeted 89Zr-Pertuzumab PET/CT. Radiology. 2020 Aug;296(2):370-378. doi: 10.1148/radiol.2020192828. Epub 2020 Jun 9. PMID 32515679
- [Derived] Ulaner GA, Hyman DM, Lyashchenko SK, Lewis JS, Carrasquillo JA. 89Zr-Trastuzumab PET/CT for Detection of Human Epidermal Growth Factor Receptor 2-Positive Metastases in Patients With Human Epidermal Growth Factor Receptor 2-Negative Primary Breast Cancer. Clin Nucl Med. 2017 Dec;42(12):912-917. doi: 10.1097/RLU.0000000000001820. PMID 28872549
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- HER2-targeted PET/CT: Pts with confirmed HER2- breast cancer will undergo HER2-targeted PET/CT. 89Zr-trastuzumab is a novel radiotracer which allows excellent visualization of HER2+ lesions. 89Zr-pertuzumab is a novel radiotracer which may allow for specific visualization of HER2+ lesions. PET/CT imaging with these novel radiotracers will allow evaluation of all identifiable malignant lesions, rather than evaluation of only single lesions by biopsy.
Period: Overall Study
Arm/Group | HER2-targeted PET/CT
Started | 49
Completed | 43
Not Completed | 6
Not completed — Not Treated | 4
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | HER2-targeted PET/CT
Number analyzed (Participants) | 49
Age, Continuous [Median (Full Range); unit: years] | 51 [38 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 44
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 36
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 49

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With HER2- Primary Breast Cancer Who Develop Imagable HER2+ Metastases
Description: Both SUVmax and SUVpeak will be recorded for lesions, and SUVmax and SUVaverage will be recorded for background measurements. Only those foci qualitatively scored conspicuously positive by both readers (scores of 4 or 5) will be considered as "positive".
Time Frame: 3 years
Population: Thirteen percent of women with HER2-negative primary malignancy has HER2-positive metastatic disease detected by HER2-targeted imaging.
Measure: Number; unit: % of participants
Arm/Group | HER2-targeted PET/CT
Number analyzed (Participants) | 49
% of participants | 13

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | HER2-targeted PET/CT
All-Cause Mortality (participants affected / at risk) | 37/49
Serious Adverse Events (participants affected / at risk) | 6/49
Other Adverse Events (participants affected / at risk) | 0/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HER2-targeted PET/CT (N=49)
Abdominal pain (Gastrointestinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Death NOS (General disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-21): https://cdn.clinicaltrials.gov/large-docs/43/NCT02286843/Prot_SAP_000.pdf